CLINICAL TRIAL: NCT07166497
Title: Evaluation of the Effect of the Product RV4660C CY0203 on Clinical, Biometrological and Biological Parameters in Adults With Mild to Moderate Atopic Dermatitis, an Exploratory Study
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV4660C20230530
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Mild to Moderate Atopic Dermatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Test Group
  Interventions: Other: Cosmetic product RV4660C CY0203

INTERVENTIONS:
Other: Cosmetic product RV4660C CY0203 — The product was applied once a day, in the evening, on the whole body/ off face on previously cleansed skin. The product was warmed in the hands before being applied in wide movements.

SUMMARY:
In this exploratory study, we assessed the efficacy of a cosmetic product in adults suffering from mild to moderate atopic dermatitis. This exploratory study has been conducted as a monocentric non randomized study.

To perform this clinical study, 21 non menopausal women, aged from 18 years and older, suffering from mild to moderate atopic dermatitis were enrolled.

The subjects applied the investigational product once a day, in the evening on the whole body/ off face for up to 31 days.

4 visits were planned:

* Visit 1 - Day 1 - Inclusion visit
* Visit 2 - Day 8 - Intermediate visit
* Visit 3 - Day 29 (± 3 days) - Intermediate visit
* Visit 4 - Day 36 (± 3 days) - End of study visit

ELIGIBILITY:
Main inclusion criteria :

* Woman 18 years or older
* Non-menopausal woman
* Subject with phototype I, II, III, IV as classified by Fitzpatrick
* Subject with AD according to "The U.K. Working Party's Diagnostic Criteria for Atopic Dermatitis"
* Mild to moderate AD with SCORAD (SCORing Atopic Dermatitis) between 20 and 40 inclusive
* Subject who had at least 1 inflammatory AD flare-up in target areas in the year prior to inclusion visit
* Subject with at least one measuring target area on each upper or lower limb and defined as a typical AD flare-up area in the opinion of the subject
* Subject with at least one target area on each upper or lower limb with the following SCORAD target signs (between 3 and 18):

  1. Erythema ≥ 1
  2. Xerosis > 1
* Subject with pruritus intensity ≥ 3 on SCORAD analog visual scale (VAS)

Main non-inclusion criteria:

* Subject with superinfected AD
* Subject with a known history of allergy or intolerance to the components of the study product
* Subject with a dermatological condition other than AD, or characteristics (for example, tattoo) on the study areas, likely to interfere with the study evaluations according to the investigator's opinion
* Subject with another dermatological condition, acute or chronic pathology, or history of pathology, likely to interfere with study evaluations, or considered dangerous to the subject or incompatible with study requirements, in the opinion of the investigator
* Topical or oral treatment established or modified during the previous weeks or planned to be established or modified during the study, liable to interfere with the evaluation of the efficacy or cutaneous tolerance of the investigational product according to the investigator's assessment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is disseminated to the database of potential subjects by email and, if needed, by telephone, describing study title,name(s), address(es) and contacts of the study site(s), name of the Principal Investigator, the parameter(s) in study, study inclusion and exclusion criteria, study objective(s), groups of treatment, namely, if experimental or comparative products are tested, potential risks of adverse events and study duration.
  The subjects that manifested interest in participating in the study might be contacted by telephone.
  Screening questions are asked in order to screen the main inclusion and exclusion criteria Subjects' answers to the telephonic recruitment are evaluated by the Principal Investigator who decides if the subject is to be selected for the recruitment visit.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Severity of atopic dermatitis throughout the body with SCORAD (SCOring Atopic Dermatitis) | Before application and before wearing the connected watch (Day 1, Visit 1), after 7 consecutive days of wearing connected watch - before application (Day 8, Visit 2), after 21 (Day 29, Visit 3) and 28 (Day 36, Visit 4) consecutive days of application
  Evaluation performed by the investigator of
  * The extent of the disease using the rule of nines to estimate percentage of the affected body surface area. The maximum value for the extent of the disease is 100%.
  * The disease intensity calculated based on six characteristics: erythema, edema, oozing/crusts, excoriations, lichenification, and dryness. Each characteristic is given a score between 0 and 3, where 0 is absent and 3 is severe. The scores for each characteristic are added together for a total intensity score of up to 18.
  Evaluation performed by the subject of subjective symptoms including sleep loss and pruritus using a 10 cm visual analogue scale with a total maximum score of 20.
  The SCORAD was then calculated with the following formula:
  Extent/5 + 7×Intensity/2 + Subjective Symptoms
Severity of the target atopic dermatitis areas (defined as a typical AD flare-up area in the opinion of the subject) with target SCORAD | Before application and before wearing the connected watch (Day 1, Visit 1), after 7 consecutive days of wearing connected watch - before application (Day 8, Visit 2), after 21 (Day 29, Visit 3) and 28 (Day 36, Visit 4) consecutive days of application
  Evaluation performed by the investigator of severity of the target areas calculated based on six characteristics: erythema, edema, oozing/crusts, excoriations, lichenification, and dryness. Each characteristic is given a score between 0 and 3, where 0 is absent and 3 is severe. The scores for each characteristic are added together for a total intensity score of up to 18.
The pruritus severity with the Chronic itch burden scale over the past 7 days | Before application and before wearing the connected watch (Day 1, Visit 1), after 7 consecutive days of wearing connected watch - before application (Day 8, Visit 2), after 21 (Day 29, Visit 3) and 28 (Day 36, Visit 4) consecutive days of application
  Evaluation performed by the subject of pruritus severity on a NRS (0=no itching to 10=worst itching imaginable) over the past 7 days
The impact of pruritus on quality of life with the Chronic itch burden scale over the past 7 days | Before application and before wearing the connected watch (Day 1, Visit 1), after 7 consecutive days of wearing connected watch - before application (Day 8, Visit 2), after 21 (Day 29, Visit 3) and 28 (Day 36, Visit 4) consecutive days of application
  Evaluation performed by the subject of the impact of pruritus on daily life over the past 7 days with 20 questions from 0=not at all, 1=a little, 2=somewhat, 3=a lot and 4=very much
The pruritus severity with VAS (Visual Analog Scale) over the last 72 hours | Before application and before wearing the connected watch (Day 1, Visit 1), after 7 consecutive days of wearing connected watch - before application (Day 8, Visit 2), after 21 (Day 29, Visit 3) and 28 (Day 36, Visit 4) consecutive days of application
  Evaluation performed by the subject of pruritus severity using a VAS (continuous sliding scale from 0 cm = no itching to 10 cm = worst itching imaginable) over the last 72 hours using the SCORAD scale
The pruritus severity with VAS (Visual Analog Scale) over the last 24 hours | Before application and before wearing the connected watch (Day 1, Visit 1), after 7 consecutive days of wearing connected watch - before application (Day 8, Visit 2), after 21 (Day 29, Visit 3) and 28 (Day 36, Visit 4) consecutive days of application
  Evaluation performed by the subject of pruritus severity using a VAS (continuous sliding scale from 0 cm = no itching to 10 cm = worst itching imaginable) over the last 24 hours
The quality of sleep using connected watch | Before products' application from Day 1 to Day 7 and after 21 consecutive days of products' application from Day 8 to Day 29.
  Measurement of sleep parameters using a connected watch worn on the wrist by the subjects
The quality of sleep with VAS (Visual Analog Scale) | Before application and before wearing the connected watch (Day 1, Visit 1), after 7 consecutive days of wearing connected watch - before application (Day 8, Visit 2), after 21 (Day 29, Visit 3) and 28 (Day 36, Visit 4) consecutive days of application
  Evaluation performed by the subject of quality of sleep using a VAS (continuous sliding scale from 0 cm = no sleep disturbance to 10 cm = worst sleep disturbance imaginable) over the last 72 hours using the SCORAD scale
The quality of sleep with the Chronic itch burden scale | Before application and before wearing the connected watch (Day 1, Visit 1), after 7 consecutive days of wearing connected watch - before application (Day 8, Visit 2), after 21 (Day 29, Visit 3) and 28 (Day 36, Visit 4) consecutive days of application
  Evaluation performed by the subject of quality of sleep using the question n°4 from the Chronic Itch Burden Scale questionnaire
The quality of sleep with the Sleep Health index | Before application and before wearing the connected watch (Day 1, Visit 1), after 7 consecutive days of wearing connected watch - before application (Day 8, Visit 2), after 21 (Day 29, Visit 3) and 28 (Day 36, Visit 4) consecutive days of application
  Evaluation performed by the subject of quality of sleep using the questions n°6 to 10 from the Sleep Health index
The quality of sleep using Insomnia Severity Index (ISI) questionnaire | Before application and before wearing the connected watch (Day 1, Visit 1), after 7 consecutive days of wearing connected watch - before application (Day 8, Visit 2), after 21 (Day 29, Visit 3) and 28 (Day 36, Visit 4) consecutive days of application
  Evaluation performed by the subject of the quality of sleep
The scratch using a connected watch | Before products' application from Day 1 to Day 7 and after 21 consecutive days of products' application from Day 8 to Day 29.
  Measurement of scratch using a connected watch worn on the wrist by the subjects
The skin hydration using a Corneometer | Before application and before wearing the connected watch (Day 1, Visit 1), after 7 consecutive days of wearing connected watch - before application (Day 8, Visit 2), after 21 (Day 29, Visit 3) and 28 (Day 36, Visit 4) consecutive days of application
  Evaluation of the hydration index performed by a clinical research technician on one of the target area
The skin barrier condition using a Vapometer | Before application and before wearing the connected watch (Day 1, Visit 1), after 7 consecutive days of wearing connected watch - before application (Day 8, Visit 2), after 21 (Day 29, Visit 3) and 28 (Day 36, Visit 4) consecutive days of application
  Evaluation of the trans-epidermal water loss performed by a clinical research technician on one of the target area
The skin microbiota with non-invasive skin swabs | Before product's application (Day 8, Visit 2) and after 28 consecutive days of product's application (Day 36, Visit 4)
  Evaluation of the skin microbiota performed by a clinical research technician on one of the target areas
Metabolites produced by host and microorganisms of the skin with non-invasive skin D-Squames | Before product's application (Day 8, Visit 2) and after 28 consecutive days of product's application (Day 36, Visit 4)
  Evaluation of the metabolites produced by host and microorganisms of the skin performed by a clinical research technician on one of the target areas
Metabolites produced by host and microorganisms of the skin with non-invasive skin swabs | Before product's application (Day 8, Visit 2) and after 28 consecutive days of product's application (Day 36, Visit 4)
  Evaluation of the metabolites produced by host and microorganisms of the skin performed by a clinical research technician on one of the target areas

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Research Center, Toulouse, France, France